CLINICAL TRIAL: NCT00408694
Title: A Phase II Study of Concurrent Chemoradiotherapy Using Three-Dimensional Conformal Radiotherapy (3D-CRT) or Intensity-Modulated Radiation Therapy (IMRT) + Bevacizumab (BV) for Locally or Regionally Advanced Nasopharyngeal Cancer
Brief Title: Bevacizumab, Cisplatin, Radiation Therapy, and Fluorouracil in Treating Patients With Stage IIB, Stage III, Stage IVA, or Stage IVB Nasopharyngeal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Radiation Therapy Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00736; NCI-2009-00736 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RTOG-0615; CDR0000518526; RTOG 0615 (Other: Radiation Therapy Oncology Group); RTOG-0615 (Other: CTEP); U10CA021661 (NIH); NCT00707096 (obsolete NCT alias)
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Results first posted 2013-04-18 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Stage II Nasopharyngeal Keratinizing Squamous Cell Carcinoma AJCC v7; Stage III Nasopharyngeal Keratinizing Squamous Cell Carcinoma AJCC v7; Stage III Nasopharyngeal Undifferentiated Carcinoma AJCC v7; Stage IV Nasopharyngeal Keratinizing Squamous Cell Carcinoma AJCC v7; Stage IV Nasopharyngeal Undifferentiated Carcinoma AJCC v7
MeSH Terms: interventions — Radiotherapy, Conformal; Bevacizumab; Immunoglobulin G; Disulfides; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Fluorouracil; dehydroftorafur; Radiotherapy, Intensity-Modulated

ARMS (1):
- Treatment (bevacizumab, cisplatin, fluorouracil, IMRT, 3D-CRT) (Experimental): BEVACIZUMAB AND CHEMORADIOTHERAPY: Patients receive bevacizumab IV over 30-90 minutes and cisplatin IV over 20-30 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Beginning in week 1, patients also undergo three-dimensional conformal radiotherapy or intensity-modulated radiotherapy once daily 5 days a week for a total of 33 fractions.
  ADJUVANT THERAPY: Beginning in week 10, patients receive fluorouracil IV continuously over 96 hours on days 1-4, cisplatin IV over 20-30 minutes on day 1 OR days 1 and 2, and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Biological: Bevacizumab; Drug: Cisplatin; Drug: Fluorouracil; Radiation: Intensity-Modulated Radiation Therapy

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3D-CRT
  Other Names: 3-dimensional radiation therapy; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; BEVACIZUMAB, LICENSE HOLDER UNSPECIFIED; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy

SUMMARY:
This phase II trial is studying how well giving bevacizumab together with cisplatin, radiation therapy, and fluorouracil works in treating patients with stage IIB, stage III, stage IVA, or stage IVB nasopharyngeal cancer. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of nasopharyngeal cancer by blocking blood flow to the tumor. Drugs used in chemotherapy, such as cisplatin and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving bevacizumab together with chemotherapy and radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and tolerability of bevacizumab and chemoradiotherapy comprising cisplatin and radiotherapy followed by adjuvant therapy comprising cisplatin, fluorouracil, and bevacizumab in patients with stage IIB-IVB nasopharyngeal cancer.

SECONDARY OBJECTIVES:

I. Determine the 1- and 2-year rates of locoregional progression-free in patients treated with this regimen.

II. Determine the 1- and 2-year rates of distant metastases-free in patients treated with this regimen.

III. Determine the 1- and 2-year rates of progression-free and overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

BEVACIZUMAB AND CHEMORADIOTHERAPY: Patients receive bevacizumab IV over 30-90 minutes and cisplatin IV over 20-30 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Beginning in week 1, patients also undergo three-dimensional conformal radiotherapy or intensity-modulated radiotherapy once daily 5 days a week for a total of 33 fractions.

ADJUVANT THERAPY: Beginning in week 10, patients receive fluorouracil IV continuously over 96 hours on days 1-4, cisplatin IV over 20-30 minutes on day 1 OR days 1 and 2, and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cancer of the nasopharynx based on biopsy of a primary lesion and/or lymph nodes

  * Histologic WHO types I-IIb/III
* Stage IIB-IVB disease

  * No T1-2, N1 disease in which node positivity is based on the presence of retropharyngeal lymph nodes
* No distant metastases
* Zubrod performance status 0-1
* WBC ? 4,000/mm?
* Hemoglobin ? 9.0 g/dL
* Platelet count ? 100,000/mm?
* Absolute neutrophil count ? 1,500/mm?
* INR ? 1.5
* aPTT ? 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ? 1.5 times ULN
* ALT and AST ? 1.5 times ULN
* Bilirubin ? 1.5 times ULN
* Creatinine ? 1.5 mg/dL OR creatinine clearance ? 55 mL/min
* Urine protein:creatinine (UPC) ratio < 1.0

  * If UPC > 0.5, 24-hour urine protein must be < 1,000 mg
* Hearing loss primarily sensorineural in nature and requiring a hearing aid or intervention that interferes in a clinically significant way with activities of daily living allowed
* Conductive hearing loss from tumor-related otitis media is allowed
* No severe, active comorbidity, including any of the following:

  * Ongoing bleeding diathesis, hemorrhagic disorder, or coagulopathy within the past 6 months
  * Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
  * Esophageal varices, nonhealing wound, nonhealing ulcer, or bone fracture within the past 6 months
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within the past 30 days
  * Unstable angina and/or congestive heart failure or peripheral vascular disease requiring hospitalization within the past 12 months
  * Major medical or psychiatric illness that, in the opinion of the study investigator, would preclude study compliance
  * Active, untreated infection and/or acute bacterial or fungal infection requiring intravenous antibiotics
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  * History of significant weight loss (> 15% from baseline)
  * History of arterial thromboembolic events
  * Acquired immune deficiency syndrome
  * Transmural myocardial infarction
  * Cerebrovascular accident
  * Transient ischemic attack
  * Any other cardiac condition that, in the opinion of the investigator, would preclude study compliance
* No gross hemoptysis or hematemesis, defined as bright red blood of ? 1 teaspoon per coughing episode, within the last 4 weeks (incidental blood mixed with phlegm allowed)
* No other invasive malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the breast, oral cavity, or cervix
* Nutritional and physical condition considered suitable for study treatment
* No significant traumatic injury within the past 4 weeks
* No history of allergic reaction to the study drugs
* No baseline blood pressure > 150/100 mm Hg
* No peripheral neuropathy ? grade 2
* Not pregnant or nursing
* Negative serum pregnancy test
* Fertile patients must use effective contraception during and for ? 6 months after completion of study treatment
* At least 10 days since prior and no concurrent dipyridamole, ticlopidine, clopidogrel bisulfate, cilostazol, warfarin, heparin, daily treatment with acetylsalicylic acid (> 325 mg/day), or nonsteroidal anti-inflammatory medications known to inhibit platelet function
* No prior head and neck surgery of the primary tumor or lymph nodes except for incisional or excisional biopsies

  * More than 15 days since prior biopsies
* More than 1 week since prior fine-needle aspirations or placement of percutaneous gastrostomy tube
* More than 4 weeks since prior major surgical procedures
* No prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* No prior bevacizumab or other vascular endothelial growth factor-targeting agents
* No prior systemic chemotherapy for the study cancer

  * Prior chemotherapy for a different cancer allowed
* No concurrent hematologic growth factors (e.g. filgrastim [G-CSF], darbepoetin alfa, epoetin alfa) during study chemoradiotherapy
* No concurrent prophylactic growth factors for neutropenia during study adjuvant therapy
* No concurrent prophylactic amifostine or pilocarpine
* No other concurrent experimental therapeutic cancer treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-12-13 (Actual); Primary Completion 2011-12-15 (Actual); Study Completion 2011-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lee, Principal Investigator — Radiation Therapy Oncology Group
Locations (108):
- United States (104):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Mercy General Hospital Radiation Oncology Center, Sacramento, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Integrated Community Oncology Network-Southside Cancer Center, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network-Florida Cancer Center Beaches, Jacksonville Beach, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - 21st Century Oncology-Orange Park, Orange Park, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - 21st Century Oncology-Palatka, Palatka, Florida
  - Integrated Community Oncology Network-Flager Cancer Center, Saint Augustine, Florida
  - Memorial University Medical Center, Savannah, Georgia
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Saint Vincent Anderson Regional Hospital/Cancer Center, Anderson, Indiana
  - Union Hospital of Cecil County, Elkton, Maryland
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Singing River Hospital, Pascagoula, Mississippi
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Beth Israel Medical Center, New York, New York
  - Saint Luke's Roosevelt Hospital Center - Saint Luke's Division, New York, New York
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - UPMC Cancer Center at Clarion Hospital, Clarion, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Upper Delaware Valley Cancer Center, Milford, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - UPMC Cancer Center-Natrona Heights, Natrona Heights, Pennsylvania
  - UPMC Jameson, New Castle, Pennsylvania
  - Radiation Therapy Oncology Group, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - AnMed Health Hospital, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - London Regional Cancer Program, London, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - McGill University Department of Oncology, Montreal, Quebec

REFERENCES:
- [Derived] Lee NY, Harris J, Kim J, Garden A, Mechalakos J, Pfister DG, Chan ATC, Hu K, Colevas AD, Frank S, Shenouda G, Bar-Ad V, Waldron JN, Harari PM, Raben A, Torres-Saavedra P, Le QT. Long-term Outcomes of Bevacizumab and Chemoradiation for Locoregionally Advanced Nasopharyngeal Carcinoma: A Nonrandomized Controlled Trial. JAMA Netw Open. 2023 Jun 1;6(6):e2316094. doi: 10.1001/jamanetworkopen.2023.16094. PMID 37266942
- [Derived] Lee NY, Zhang Q, Pfister DG, Kim J, Garden AS, Mechalakos J, Hu K, Le QT, Colevas AD, Glisson BS, Chan AT, Ang KK. Addition of bevacizumab to standard chemoradiation for locoregionally advanced nasopharyngeal carcinoma (RTOG 0615): a phase 2 multi-institutional trial. Lancet Oncol. 2012 Feb;13(2):172-80. doi: 10.1016/S1470-2045(11)70303-5. Epub 2011 Dec 15. PMID 22178121

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Bevacizumab, Cisplatin, Fluorouracil, IMRT, 3D-CRT): BEVACIZUMAB AND CHEMORADIOTHERAPY: Patients receive bevacizumab IV over 30-90 minutes and cisplatin IV over 20-30 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Beginning in week 1, patients also undergo three-dimensional conformal radiotherapy or intensity-modulated radiotherapy once daily 5 days a week for a total of 33 fractions.
  ADJUVANT THERAPY: Beginning in week 10, patients receive fluorouracil IV continuously over 96 hours on days 1-4, cisplatin IV over 20-30 minutes on day 1, and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Bevacizumab, Cisplatin, Fluorouracil, IMRT, 3D-CRT)
Started | 46
Completed | 44 (Subjects contributing data to the primary analysis are considered to have completed the study.)
Not Completed | 2
Not completed — Ineligible | 1
Not completed — No protocol treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Bevacizumab, Cisplatin, Fluorouracil, IMRT, 3D-CRT)
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 48 [18 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a Grade 4 Hemorrhage or Any Grade 5 Adverse Event Assessed to be Definitely, Probably, or Possibly Related to Protocol Treatment During the First Year.
Description: Estimated using a binomial distribution along with the 95% confidence interval. Adverse events (AE) are graded using CTCAE v3.0. Grade refers to the severity of the AE. The CTCAE v3.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE.
Time Frame: From start of treatment to one year.
Population: Eligible patients who started study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Bevacizumab, Cisplatin, Fluorouracil, IMRT, 3D-CRT)
Number analyzed (Participants) | 44
percentage of participants | 0 [0 to 0]
Statistical Analysis 1: Comparison: Treatment (Bevacizumab, Cisplatin, Fluorouracil, IMRT, 3D-CRT); Null hypothesis, H0: Incidence of patients with either grade 4 hemorrhage or any grade 5 adverse event for the protocol treatment regimen ≤ 0.05. Alternative hypothesis, HA: Incidence of patients with either grade 4 hemorrhage or any grade 5 adverse event for the protocol treatment regimen ≥ 0.15; Test type: Other; If 3 of the first 14 patients or 4 of the first 42 patients experience the specified adverse events, then the regimen is considered unacceptable as calculated by the Fleming method for a two-stage design with type I error and the statistical power were set at 0.14 and 0.83, respectively

2. Secondary Outcome: Percentage of Patients With Grade 4 Hemorrhage or Any Grade 5 Adverse Event Assessed to be Definitely, Probably, or Possibly Related to Protocol Treatment After the First Year.
Description: as for outcome 1
Time Frame: Analysis occurs after all patients have been on study for at least 2 years. Patients are followed from day 366 to death or study termination whichever occurs first, up to 3.6 years.
Population: Eligible patients who started study treatment and survived more than one year.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Bevacizumab, Cisplatin, Fluorouracil, IMRT, 3D-CRT)
Number analyzed (Participants) | 41
percentage of participants | 0 [0 to 0]

3. Secondary Outcome: Patient Tolerability to Each Component (Concurrent and Adjuvant) of the Protocol Treatment Regimen
Description: Evaluated in terms of protocol treatment delivery. For concurrent treatment, measured by the percentage of patients who received 2 or more cycles of cisplatin (CDDP) and bevacizumab (BV) during concurrent treatment with radiation therapy(RT) and who had RT scored by the study chair as no variation or minor variation. For adjuvant treatment, measured by the percentage of patients who received 2 or more cycles of CDDP and 5-FU and BV during the adjuvant treatment phase. Estimated using a binomial distribution along with their associated 95% confidence intervals.
Time Frame: From start of treatment to end of treatment (approximately day 109).
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Bevacizumab, Cisplatin, Fluorouracil, IMRT, 3D-CRT)
Number analyzed (Participants) | 44
percentage of participants
  Concurrent component | 68.2 [52.4 to 81.4]
  Adjuvant component | 68.2 [52.4 to 81.4]

4. Secondary Outcome: Death During or Within 30 Days of Discontinuation of Protocol Treatment.
Description: The percentage of patients dying during protocol treatment or within 30 days after the end of treatment. Estimated using a binomial distribution along with associated 95% confidence interval.
Time Frame: From start of treatment to 30 days after end of treatment (treatment ends approximately day 109).
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Bevacizumab, Cisplatin, Fluorouracil, IMRT, 3D-CRT)
Number analyzed (Participants) | 44
percentage of participants | 0 [0 to 0]

5. Secondary Outcome: One- and Two-year Distant Metastases-free Rates
Description: Distant metastasis is defined as clear evidence of distant metastases (lung, bone, brain, etc.); biopsy is recommended where possible. Distant metastasis-free rate estimated by cumulative incidence method with death considered a competing risk.
Time Frame: From registration to two years
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Bevacizumab, Cisplatin, Fluorouracil, IMRT, 3D-CRT)
Number analyzed (Participants) | 44
percentage of participants
  One-year | 97.7 [93.3 to 100.0]
  Two-year | 90.8 [82.2 to 99.5]

6. Secondary Outcome: One- and Two-year Loco-regional Progression-free Rates
Description: Loco-regional progression is defined as an estimated increase in the size of the tumor (product of the perpendicular diameters of the two largest dimensions) of greater than 25%, taking as reference the smallest value of all previous measurements or appearance of new areas of malignant disease. Local-regional progression-free rate estimated by cumulative incidence with death considered a competing risk.
Time Frame: Analysis occurs after all patients have been on study for at least 2 years. Patients are followed from study registration to death or study termination whichever occurs first, up to 3.6 years.
Population: Eligible patients who started study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Bevacizumab, Cisplatin, Fluorouracil, IMRT, 3D-CRT)
Number analyzed (Participants) | 44
percentage of participants
  One-year | 93.2 [85.6 to 100.0]
  Two-year | 74.7 [61.8 to 87.6]

7. Secondary Outcome: One- and Two-year Progression-free Survival Rates
Description: Progression-free survival rate estimated by Kaplan-Meier method along with 95% confidence interval. An event is loco-regional or distant progression, or death due to any cause. Loco-regional progression is defined as an estimated increase in the size of the tumor (product of the perpendicular diameters of the two largest dimensions) of greater than 25%, taking as reference the smallest value of all previous measurements or appearance of new areas of malignant disease. Distant progression is defined as distant metastases.
Time Frame: as for outcome 6
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Bevacizumab, Cisplatin, Fluorouracil, IMRT, 3D-CRT)
Number analyzed (Participants) | 44
percentage of participants
  One-year | 90.9 [82.4 to 99.4]
  Two-year | 74.7 [61.8 to 87.6]

8. Secondary Outcome: One- and Two-year Overall Survival Rates
Description: Overall survival rate estimated by Kaplan-Meier method along with 95% confidence interval. An event is death due to any cause.
Time Frame: as for outcome 6
Population: Eligible patients who started study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Bevacizumab, Cisplatin, Fluorouracil, IMRT, 3D-CRT)
Number analyzed (Participants) | 44
percentage of participants
  One-year | 93.2 [85.7 to 100.0]
  Two-year | 90.9 [82.3 to 99.4]

9. Secondary Outcome: Percentage of Patients With Other Grade 3-5 Adverse Events Assessed to be Definitely, Probably, or Possibly Related to Protocol Treatment
Description: as for outcome 1
Time Frame: Analysis occurs after all patients have been on study for at least 2 years. Patients are followed from start of treatment to death or study termination whichever occurs first, up to 3.6 years.
Population: Eligible patients who started treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Bevacizumab, Cisplatin, Fluorouracil, IMRT, 3D-CRT)
Number analyzed (Participants) | 44
percentage of participants | 90.9 [78.3 to 97.5]

ADVERSE EVENTS:
Description: Per the protocol, toxicity was collected via CTCAE 3.0 then mapped to CTCAE 4.0 for reporting on this website. Subjects experiencing more than one of a given adverse event (AE) are counted only once for that AE.
Groups:
- Treatment (Bevacizumab, Cisplatin, Fluorouracil, IMRT, 3D-CRT): BEVACIZUMAB AND CHEMORADIOTHERAPY: Patients receive bevacizumab IV over 30-90 minutes and cisplatin IV over 20-30 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Beginning in week 1, patients also undergo three-dimensional conformal radiotherapy or intensity-modulated radiotherapy once daily 5 days a week for a total of 33 fractions.
  ADJUVANT THERAPY: Beginning in week 10, patients receive fluorouracil IV continuously over 96 hours on days 1-4, cisplatin IV over 20-30 minutes on day 1, and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  Data is reported for eligible patients with adverse event data who started study treatment, which is 44 patients.
Arm/Group | Treatment (Bevacizumab, Cisplatin, Fluorouracil, IMRT, 3D-CRT)
Serious Adverse Events (participants affected / at risk) | 28/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Bevacizumab, Cisplatin, Fluorouracil, IMRT, 3D-CRT) (N=44)
Anemia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Paroxysmal atrial tachycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 3
Conjunctivitis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 6
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 7
Oral pain (Gastrointestinal disorders) | 2
Rectal fistula (Gastrointestinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Chills (General disorders) | 1
Fatigue (General disorders) | 5
Fever (General disorders) | 3
General disorders and administration site conditions - Other (General disorders) | 1
Catheter related infection (Infections and infestations) | 1
Infections and infestations - Other (Infections and infestations) | 5
Lung infection (Infections and infestations) | 1
Penile infection (Infections and infestations) | 1
Peripheral nerve infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood antidiuretic hormone abnormal (Investigations) | 1
Lymphocyte count decreased (Investigations) | 2
Neutrophil count decreased (Investigations) | 6
Platelet count decreased (Investigations) | 4
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 5
Acidosis (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 9
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 4
Erectile dysfunction (Reproductive system and breast disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Hypertension (Vascular disorders) | 3
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Bevacizumab, Cisplatin, Fluorouracil, IMRT, 3D-CRT) (N=44)
Anemia (Blood and lymphatic system disorders) | 18
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Hemolysis (Blood and lymphatic system disorders) | 2
Paroxysmal atrial tachycardia (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 2
External ear inflammation (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 20
Middle ear inflammation (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 14
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 4
Blurred vision (Eye disorders) | 1
Eye disorders - Other (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Anal mucositis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 22
Dental caries (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 10
Dry mouth (Gastrointestinal disorders) | 42
Dyspepsia (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 42
Esophageal pain (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 3
Lip pain (Gastrointestinal disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 40
Nausea (Gastrointestinal disorders) | 32
Oral pain (Gastrointestinal disorders) | 14
Rectal fistula (Gastrointestinal disorders) | 1
Rectal pain (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 21
Chills (General disorders) | 4
Edema face (General disorders) | 10
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 35
Fever (General disorders) | 11
General disorders and administration site conditions - Other (General disorders) | 2
Pain (General disorders) | 9
Allergic reaction (Immune system disorders) | 1
Gum infection (Infections and infestations) | 4
Infections and infestations - Other (Infections and infestations) | 8
Lung infection (Infections and infestations) | 2
Peripheral nerve infection (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 22
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 20
Activated partial thromboplastin time prolonged (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 5
Blood bilirubin increased (Investigations) | 3
Creatinine increased (Investigations) | 7
GGT increased (Investigations) | 1
INR increased (Investigations) | 2
Investigations - Other (Investigations) | 4
Lymphocyte count decreased (Investigations) | 9
Neutrophil count decreased (Investigations) | 14
Platelet count decreased (Investigations) | 13
Weight loss (Investigations) | 19
White blood cell decreased (Investigations) | 17
Acidosis (Metabolism and nutrition disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 12
Dehydration (Metabolism and nutrition disorders) | 10
Hyperglycemia (Metabolism and nutrition disorders) | 14
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 14
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypokalemia (Metabolism and nutrition disorders) | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 10
Hyponatremia (Metabolism and nutrition disorders) | 15
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Trismus (Musculoskeletal and connective tissue disorders) | 15
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Accessory nerve disorder (Nervous system disorders) | 1
Acoustic nerve disorder NOS (Nervous system disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 23
Dysphasia (Nervous system disorders) | 1
Extrapyramidal disorder (Nervous system disorders) | 1
Facial muscle weakness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 10
Myelitis (Nervous system disorders) | 4
Nervous system disorders - Other (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 16
Peripheral motor neuropathy (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 24
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 6
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 7
Insomnia (Psychiatric disorders) | 4
Psychosis (Psychiatric disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 1
Irregular menstruation (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 10
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 8
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 24
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 11
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 13
Alopecia (Skin and subcutaneous tissue disorders) | 15
Dry skin (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Skin atrophy (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 12
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Skin induration (Skin and subcutaneous tissue disorders) | 20
Flushing (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 2
Hypertension (Vascular disorders) | 5
Lymphedema (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less